CLINICAL TRIAL: NCT03962504
Title: An Efficient, Exposure-based Treatment for PTSD Compared to Prolonged Exposure: A Non-inferiority Randomized Trial
Brief Title: Written Exposure Therapy Versus Prolonged Exposure: a Non-inferiority Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MHBB-005-18F; CX001967-01 (Other Grant/Funding Number: Department of Veterans Affairs)
Record Dates: First submitted 2019-05-22; First posted 2019-05-24 (Actual); Results first posted 2024-07-18 (Actual); Last update posted 2024-07-18 (Actual); Status verified 2024-04

CONDITIONS: PTSD
Keywords: PTSD; psychosocial treatment; cognitive behavioral treatment; veterans; quality of life
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: The study is a non-inferiority design to examine if a brief intervention for PTSD is non-inferior to a more time-intensive intervention.
Who Masked: Outcomes Assessor
Masking Description: Assessors will be unaware of participant conditions. Assessors will not have access to any study materials in which unmasking could occur. Participants will be instructed to not reveal their treatment condition to the assessors.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- written exposure therapy (Experimental): The WET condition consists of 5-7 weekly treatment sessions, with the first session lasting 1 hour and each subsequent session lasting approximately 40 minutes. The first session consists of education about common trauma reactions and the WET rationale. The participant is then given general instructions for completing the trauma narratives and specific instructions for completing the first 30-minute narrative writing session. All WET sessions begin with the therapist reading the specific writing instructions, clarifying any questions the person has, and leaving the instructions with the participant during the 30-minute writing session. Writing instructions begin with a focus on the details of the trauma and then shift to the meaning of the trauma event. After 30 minutes of writing, the therapist stops the writing and conducts a 5-10 minute check-in regarding how the writing session went for the participant.
  Interventions: Behavioral: trauma-focused treatment
- Prolonged Exposure (Active Comparator): Prolonged Exposure (PE) is a 8-15, 90 minute trauma-focused treatment which consists of imaginal and in vivo exposures
  Interventions: Behavioral: trauma-focused treatment

INTERVENTIONS:
Behavioral: trauma-focused treatment — cognitive behavioral treatment for posttraumatic stress disorder that consists of exposure to the trauma memory.

SUMMARY:
The goal of this study is to examine whether a brief, exposure-based treatment (Written Exposure Therapy) approach is just as effective in the treatment of posttraumatic stress disorder (PTSD) compared with a more commonly used time-intensive approach called Prolonged Exposure. One hundred and fifty Veterans diagnosed with PTSD will be randomly assigned to either Written Exposure therapy or Prolonged Exposure. Veteran participants will be assessed at pre-treatment, and 10-, 20-, and 30- weeks post first treatment session. Primary outcome measure will be PTSD symptom severity. The secondary outcome measure will be quality of life. In addition, treatment dropout during the first five sessions will be examined. WET is expected to have a lower treatment dropout rate relative to PE.

DETAILED DESCRIPTION:
Although Written Exposure Therapy (WET) is listed in the upcoming VA/DoD PTSD Practice Guidelines as an evidence-based, recommended PTSD treatment, there are limited data supporting the use of WET with Veterans suffering from PTSD. Additional research is needed to support the use of WET for the treatment of Veterans diagnosed with PTSD. The goal of this study is to investigate whether WET is non-inferior in the treatment of PTSD in a sample of Veterans diagnosed with PTSD. Men and women Veterans diagnosed with PTSD will be randomly assigned to either WET (n = 88) or Prolonged Exposure (PE; n = 90). PTSD symptom severity will serve as the primary outcome. Quality of life will serve as a secondary outcome measure. Assessments will be conducted by independent evaluators at baseline, 10-, 20-, and 20-week post first treatment session. WET is expected to be non-inferior to PE in reducing PTSD symptom severity and functioning. In addition, WET is expected to have significantly lower treatment dropout rate relative to the first five sessions of PE (i.e., better treatment engagement). If WET is found to be non-inferior to the more time intensive PE treatment then the VA will have evidence to support the use of a brief PTSD treatment, which will assist in addressing the high demand for PTSD clinical services.

ELIGIBILITY:
Inclusion Criteria:

* Veteran status
* Current DSM-5 diagnosis of PTSD (assessed with the Clinician Administered PTSD Scale for DSM-5; CAPS-5)
* If taking psychotropic medication, on a stable dose for at least 30 days prior to study entry

Exclusion Criteria:

* Current engagement psychosocial treatment for PTSD
* Current diagnosis of substance dependence

  * abuse will not be excluded; determined with severe combined immunodeficiency (SCID)
* Current psychosis or unstable bipolar disorder diagnosis

  * determined with the Mini International Neuropsychiatric Interview (MINI)clinician-administered interview
* High suicidal risk

  * i.e., intent with a plan; assessed with the MINI suicide module
* Significant cognitive impairment (assessed with the Montreal Cognitive Assessment [MoCA] and clinical judgment)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 178 (Actual)
Dates: Start 2019-09-09 (Actual); Primary Completion 2023-01-02 (Actual); Study Completion 2023-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Denise M Sloan, PhD, Principal Investigator — VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA
Locations (3):
- United States (3):
  - VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA, Boston, Massachusetts
  - Ralph H. Johnson VA Medical Center, Charleston, SC, Charleston, South Carolina
  - William S. Middleton Memorial Veterans Hospital, Madison, WI, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Datasets meeting VA standards for disclosure to the public will be made available within 1 year after publication. Prior to distribution, a local privacy officer will certify that all datasets contains no protected health information (PHI). Final data sets will be maintained locally until enterprise-level resources become available for long-term storage and access. Guidance on request and distribution processes will be provided by Office of Research and Development (ORD). Those requesting data will be asked to sign a Letter of Agreement.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: one year

REFERENCES:
- [Derived] Sloan DM, Marx BP, Acierno R, Messina M, Muzzy W, Gallagher MW, Litwack S, Sloan C. Written Exposure Therapy vs Prolonged Exposure Therapy in the Treatment of Posttraumatic Stress Disorder: A Randomized Clinical Trial. JAMA Psychiatry. 2023 Nov 1;80(11):1093-1100. doi: 10.1001/jamapsychiatry.2023.2810. PMID 37610727

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Written Exposure Therapy | Prolonged Exposure
Started | 88 | 90
Completed | 77 | 58
Not Completed | 11 | 32
Not completed — Other | 11 | 32

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Written Exposure Therapy | Prolonged Exposure | Total
Number analyzed (Participants) | 88 | 90 | 178
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.17 (13.33) | 43.79 (13.96) | 44.97 (13.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 23 | 44
  Male | 67 | 67 | 134
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 2 | 5
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 3 | 1 | 4
  Black or African American | 19 | 15 | 34
  White | 55 | 54 | 109
  More than one race | 4 | 9 | 13
  Unknown or Not Reported | 4 | 9 | 13
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 88 | 90 | 178

OUTCOME MEASURES:

1. Primary Outcome: Clinician Administered PTSD Scale for Diagnostic (CAPS-5) and Statistical Manual of Mental Disorders (DSM-5)
Description: The CAPS-5 is a structured diagnostic interview and the gold standard for assessing the DSM-5 symptoms of PTSD (American Psychiatric Association, 2013). The scale also assesses social and occupational functioning, dissociation symptoms, and the validity of symptom reports. The CAPS-5 uses a single 5-point ordinal rating scale to measure symptom severity. Symptom severity ratings combine information about symptom frequency and intensity obtained by the interviewer. Psychometric properties indicate high criterion and construct validity and high agreement with a self-report measure of PTSD (Weathers et al., 2018). The CAPS-5 requires approximately 40 minutes to administer.
  Scores can range from 0-80, with higher scores indicating greater severity.
Time Frame: change score baseline to 20 weeks
Measure: Mean (95% Confidence Interval); unit: CAPS-5 total score
Arm/Group | Written Exposure Therapy | Prolonged Exposure
Number analyzed (Participants) | 88 | 90
CAPS-5 total score | 26.17 [23.88 to 28.46] | 24.78 [22.29 to 27.27]

2. Secondary Outcome: World Health Organization Quality of Life BREF
Description: The World Health Organization Quality of Life BREF (WHOQOL-BREF; WHO, 1998) instrument comprises 26 items, which measure the following broad domains: physical health, psychological health, social relationships, and environment. The WHOQOL-BREF is a shorter version of the original instrument that is more convenient for use in large research studies or clinical trials. This measure requires 5-10 minutes to complete.
  Total score 0-100, with higher scores indicate greater quality of life.
Time Frame: change score baseline to 20 weeks
Population: The sample size is substantially less than the number randomized because the self-report measure was mailed to the study team due to COVID-19 pandemic and response rate for self-report measures was much lower than clinician-administered interviews (i.e., CAPS-5). Accordingly, the planned analysis is not conducted as it is underpowered.
Measure: Mean (Standard Deviation); unit: change score; score on a scale
Arm/Group | Written Exposure Therapy | Prolonged Exposure
Number analyzed (Participants) | 38 | 36
change score; score on a scale | 3.21 (0.49) | 4.13 (1.15)

ADVERSE EVENTS:
Time Frame: 30 weeks
Arm/Group | Written Exposure Therapy | Prolonged Exposure
All-Cause Mortality (participants affected / at risk) | 0/88 | 0/90
Serious Adverse Events (participants affected / at risk) | 4/88 | 7/90
Other Adverse Events (participants affected / at risk) | 6/88 | 5/90
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Written Exposure Therapy (N=88) | Prolonged Exposure (N=90)
medical hospitalization (Surgical and medical procedures) | 3 (3) | 3 (3) — hospitalization due to medical surgery unrelated to study
medical hospitalization (Infections and infestations) | 1 (1) | 1 (1) — hospitalized due to severe dehydration due to vomiting during flu.
psychiatric hospitalization (Psychiatric disorders) | 0 (0) | 3 (3) — increased suicidal risk
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Written Exposure Therapy (N=88) | Prolonged Exposure (N=90)
contracted COVID-19 (Immune system disorders) | 6 (6) | 5 (5) — physical symptoms from contracting COVID-19

LIMITATIONS AND CAVEATS:
Study focused on veteran participants and thus findings may not generalize to the general population. The study also primarily took place during COVID-19 global pandemic, including the height of the initial lockdown, which was a period of increased stress and anxiety.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-12-28): https://cdn.clinicaltrials.gov/large-docs/04/NCT03962504/Prot_SAP_001.pdf
  • Informed Consent Form (2021-10-18): https://cdn.clinicaltrials.gov/large-docs/04/NCT03962504/ICF_000.pdf